CLINICAL TRIAL: NCT04708899
Title: Development of an Arabic Central Auditory Processing Remediation Program for Dyslexic Children With(Central) Auditory Processing Disorder
Brief Title: Development of an Arabic Central Auditory Processing Remediation Program for Dyslexic Children With(C)APD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rana ElShafaei (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Rana ElShafaei, assistant lecturer of Phoniatrics (otorhinolaryngology department), Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00018699
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Central Auditory Processing Disorder; Dyslexia
MeSH Terms: conditions — Language Development Disorders; Dyslexia

STUDY DESIGN:
Intervention Model Description: Rehabilitation of dyslexic children with (cental) auditory processing disorder.
  The first group will receive the proposed program the arabic version of differential processing training program and the control group will receive the computer based auditory traing program (CBAT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator): cases will receive the proposed program(the arabic version of differential processing training program)
  Interventions: Behavioral: arabic version of differential processing training program
- control (Active Comparator): controls will receive the computer based auditory training program (CBAT)
  Interventions: Behavioral: Arabic computer based auditory traing program(CBAT)

INTERVENTIONS:
Behavioral: arabic version of differential processing training program — comprehensive training program for central auditory processing disorder contains auditory and linguistic tasks (language organization, phonemic and phonetic awareness, dichotic listening,temporal patterning and auditory discrimination).
  Arms: Cases
Behavioral: Arabic computer based auditory traing program(CBAT) — comprehensive computer based traing program for central auditory processing disorder contains auditory memory, temporal processing, dichotic listening , selective attention and phonemic awareness games.
  Arms: control

SUMMARY:
Rehabilitation of dyslexic children with (cental) auditory processing disorder.

The first group will receive the proposed program the arabic version of differential processing training program and the control group will receive the computer based auditory traing program (CBAT).

DETAILED DESCRIPTION:
Central Auditory Processing Disorder(C)APD is defined as difficulty for children with normal hearing to listen selectively in the presence of noise, to combine information from two ears properly, to process speech when it is slightly degraded, and to integrate auditory information when it is delivered faster than the individual with (C)APD can process.( The estimated prevalence of (C)APD in the school-aged population is approximately 2 to 5 %, and the estimated prevalence of (C)APD in the older adult population is 76 %. These percentages are higher than those affected by hearing loss.

Dyslexia and (C)APD are common comorbidities and since there is limited research on (C)APD within each related academic discipline. Furthermore the language, audiologiological , and cognitive nature of the disorder confirmed that a multi-disciplinary effort is needed in order to provide clinical decision and effective intervention for the (C)APD population. Hence Development of additional intervention tools for use in clinics, schools and home settings is warranted .

The aim of this work is to develop a novel Arabic (C)APD remediation program ,to study the outcome of the program and to validate it's effectiveness by comparing it to the Arabic computer based auditory training(CBAT) program.

ELIGIBILITY:
Inclusion Criteria:

1. dyslexic children with (C)APD
2. Age from 6-12 years.
3. No gender limit.
4. Normal peripheral hearing i.e pure tone averages (average threshold from 250to 8000 Hz) should be less than or equal 25dB hearing level bilaterally.
5. Normal speech audiometry results.
6. Normal results on immitancemetry.
7. Average or below average IQ.
8. Normal language development.

Exclusion Criteria:

1. ADHD subjects. 2. Associated neurological and psychiatric disorders.

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Effect on dichotic listening | within 6 months
  assessed by screening and full version dichotic digits test pretherapy and post therapy
Effect on speech discrimination in noise. | Within 6 months
  assesed by screening and full version(auditory figure ground) SPIN test pretherapy and post therapy
Effect on temporal processing | within 6 months
  assessed by screening and full version pitch pattern sequence test (PPST) pretherapy and post therapy

SECONDARY OUTCOMES:
change in phonological processing and awareness skills | within 6month to 1 year
  assessed by phonological awareness assessment pretherapy and post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hesham kozou, Professor, Study Chair — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No
The IPD sharing is denied due to subject confidentially issues.